CLINICAL TRIAL: NCT04490603
Title: The Effect of Virtual Reality Experience on Infusion-related Pain With Lumbar Epidural Catheterization: A Prospective, Randomized Comparative Study.
Brief Title: The Effect of Virtual Reality Experience on Infusion-related Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University (Other)
Responsible Party: Principal Investigator, Jeeyoun Moon, Associate professor, Seoul National University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2005-086-1123
Record Dates: First submitted 2020-07-26; First posted 2020-07-29 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Virtual Reality

STUDY DESIGN:
Intervention Model Description: Prospective randomized open-label clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional group (No Intervention): Drug is injected to epidural space for a total of 50 minutes. The drug injection is provided in the same way as the conventional method of injecting drugs in Seoul National University Hospital Pain Center.
- VR group (Experimental): Drug is injected to epidural space for a total of 50 minutes. The drug injection is provided with virtual reality experience. Conditions are the same in both arms except for virtual reality experience.
  Interventions: Behavioral: Virtual reality experience

INTERVENTIONS:
Behavioral: Virtual reality experience — Patients are to experice virtual reality with virtual reality experience equipment (headsets, headphones, smartphones) and virtual reality experience programs. The equipments and programs are commercialized products on the market rather than medical products.
  Arms: VR group

SUMMARY:
This clinical trial aims to analyze the effect of virtual reality experience on infusion-related pain with lumbar epidural catheterization.

DETAILED DESCRIPTION:
Patients with chronic pain are to suffer from acute pain during their chronic pain-relieving interventions. However, there is no active countermeasure against pain during these procedures. This prospective randomized clinical study seeks to find an appropriate solution to the procedure related acute pain of these patients by actively utilizing virtual reality experiences.

ELIGIBILITY:
Inclusion Criteria: If all of the following conditions are met

* A person with chronic low back pain that lasts more than 3 months due to spinal stenosis or lumbar disc disease.
* Adults over 20
* Those who decided to participate out of his/her own free will and signed in written consent

Exclusion Criteria: If the patient meets one or more of the following criteria, He or She cannot participate this clinical trial.

* In case of contraindication to general lumbar catheterization (e.g. coatulopathy, infection, etc)
* Hearing and vision impairments
* Affective disorder
* History of epilepsy or seizure
* If communication is not possible due to impaired cognitive ability
* Those who have been deemed inappropriate by the researchers

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2020-08-19 (Actual); Primary Completion 2024-12-28 (Estimated); Study Completion 2024-12-28 (Estimated)

PRIMARY OUTCOMES:
Procedure-related pain | Right after the produre for 50 minutes ended.
  Pain by NRS(Numeric rating scale): from 0(no pain) to 10(worst pain possible)

SECONDARY OUTCOMES:
Patient satisfaction with virtual reality experience | Right after the produre for 50 minutes ended.
  5-point Likert-like verbal rating scale: 1, extremely satisfied; 2, satisfied; 3, undecided; 4, dissatisfied; 5, extremely dissatisfied
Intervention-related wellness index-1 (IWI-1) | Right after the produre for 50 minutes ended.
  Drug injection-related pain (Pain by NRS(Numeric rating scale): from 0(no pain) to 10(worst pain possible)) and patient satisfaction (satisfaction score) are calculated through principal component analysis as a new variable, IW index-1 (IWI-1).
Intervention-related wellness index-2 (IWI-2) | Right after the produre for 50 minutes ended.
  Calculated as IWI-2 by summing the procedure-related pain (Pain by NRS(Numeric rating scale): from 0(no pain) to 10(worst pain possible)) and patient satisfaction (satisfaction score)

CONTACTS AND LOCATIONS:
Overall Officials: Jee Youn Moon, PhD, Study Director — Associate Professor
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No